CLINICAL TRIAL: NCT07218029
Title: An Open-label Long-term Follow-up Study to Evaluate the Effects of Sotatercept When Added to Background Pulmonary Arterial Hypertension (PAH) Therapy for the Treatment of PAH (MK-7962-038)
Brief Title: A Clinical Study of Sotatercept (MK-7962) in People With Pulmonary Arterial Hypertension (MK-7962-038)
Acronym: SOTERIA
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7962-038; 2025-521970-33-00 (Registry Identifier: EU CT); U1111-1321-4943 (Registry Identifier: UTN); MK-7962-038 (Other: MSD); MK-7962-004 (Other: MSD Obsolete Identifier); NCT04796337 (obsolete NCT alias)
Record Dates: First submitted 2025-10-07; First posted 2025-10-20 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — ACE-011

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Sotatercept (Experimental): Participants enrolling from blinded PAH sotatercept studies will begin sotatercept at a dose of 0.3 mg/kg subcutaneous (SC) injection and can titrate up to the target dose of 0.7 mg/kg SC injection for the remainder of the study. Participants enrolling from unblinded PAH sotatercept studies will continue sotatercept at their current dose and, if at a dose <0.7 mg/kg, can titrate up to the target dose of 0.7 mg/kg SC injection for the remainder of the study.
  Interventions: Biological: Sotatercept

INTERVENTIONS:
Biological: Sotatercept — Sotatercept SC injection every 3 weeks
  Other Names: MK-7962; ACE-011; ActRIIA-IgG1Fc; WINREVAIR®

SUMMARY:
Researchers are looking for more ways to treat PAH. In PAH, the blood vessels in the lungs become thick and narrow, which makes it harder for blood to flow. This causes high blood pressure in the lungs and overworks the heart. PAH can make it hard to breathe and be active. Some standard (usual) treatments for PAH can treat symptoms of PAH but do not stop PAH from getting worse.

Sotatercept is a study medicine designed to treat PAH. It is a targeted therapy, which is a treatment that works on certain proteins that play a role in causing PAH.

This is a long-term follow-up (LTFU) study. People who took part in certain other studies testing sotatercept for PAH may be able to join this study. The goal of this study is to learn about the long-term safety of sotatercept and if people tolerate it when taken with standard PAH treatment over a longer period of time.

DETAILED DESCRIPTION:
LTFU PAH sotatercept study MK-7962-004 (Obsolete Identifier: NCT04796337) has been incorporated into the current MK-7962-038 (NCT07218029) study for administrative reasons. The MK-7962-004 study is no longer enrolling participants and will be formally closed. Only those who participated in MK-7962-004 may be eligible to continue into MK-7962-038.

ELIGIBILITY:
Inclusion Criteria:

The main inclusion criteria include but are not limited to the following:

* Has completed their current respective PAH sotatercept clinical study and its requirements, and must not have discontinued early
* Is willing to adhere to the study visit schedule, and understands and will comply with all protocol requirements
* Must have the ability to understand and provide documented informed consent

Exclusion Criteria:

The main exclusion criteria include but are not limited to the following:

* Did not participate in a sotatercept PAH parent study
* Missed more than the equivalent of 4 consecutive doses between the end of parent study and the start of this study.
* Presence of an ongoing serious adverse event that occurred during a PAH sotatercept clinical study that is assessed to be possibly or probably related to sotatercept
* Is a female who is pregnant or breastfeeding
* Is or has an immediate family member who is investigational site or Sponsor staff directly involved with this study
* Is currently enrolled in another investigational product study other than a sotatercept study
* Is incapacitated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 815 (Estimated)
Dates: Start 2021-05-12 (Actual); Primary Completion 2028-12-07 (Estimated); Study Completion 2028-12-07 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Who Experience an Adverse Event (AE) | Up to approximately 90 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who experience an AE will be reported.
Number of Participants Who Discontinue Study Treatment Due to an AE | Up to approximately 86 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who discontinue study treatment due to an AE will be reported.
Number of Participants with Detectable Anti-Drug Antibodies (ADAs) | Up to approximately 88 months
  ADAs will be detected in serum. The number of participants with detectable ADAs will be reported.
Laboratory parameters (Hematology): Concentration of Platelets and Hemoglobin | Up to approximately 88 months
  Blood samples will be collected to determine the concentration of platelets and hemoglobin.
Laboratory parameters (Chemistry): Concentration of Creatinine, Total Bilirubin, and Alanine Aminotransferase (ALT) | Up to approximately 86 months
  Blood samples will be collected to determine the concentration of creatinine, total bilirubin, and ALT.
Change From Baseline in Body Weight | Baseline and up to approximately 86 months
  Change from baseline in body weight will be reported.
Change From Baseline in Blood Pressure | Baseline and up to approximately 86 months
  Change from baseline in systolic and diastolic blood pressure will be reported.
Change From Baseline in Electrocardiogram (ECG) | Baseline and up to approximately 86 months
  Change from baseline in ECG (12-lead) for the determination of Fridericia's corrected QT interval (QTcF) will be reported.

SECONDARY OUTCOMES:
Change From Baseline in 6-Minute Walk Distance (6MWD) | Baseline and up to approximately 48 months
  The 6MWD is the distance walked in 6 minutes as a measure of functional capacity. The change from baseline in 6MWD will be reported.
Change From Baseline in N-Terminal Pro-Hormone B-type Natriuretic Peptide (NT-proBNP) Levels | Baseline and up to approximately 48 months
  NT-proBNP is a circulating biomarker that reﬂects myocardial stretch. The change from baseline in NT-proBNP levels will be reported.
Change From Baseline in the Percentage of Participants Who Improve or Show Maintenance in Modiﬁed New York Heart Association/ World Health Organization Classiﬁcation of Functional Status (WHO FC) | Baseline and up to approximately 48 months
  The severity of participant's PAH symptoms will be graded using the WHO FC system. WHO functional classiﬁcation for PAH ranges from Class I (no limitation in physical activity, no dyspnea with normal activity), Class II (slight limitation of physical activity), Class III (marked limitation of physical activity) and Class IV (cannot perform physical activity without any symptoms, dyspnea at rest). Participants will be classiﬁed as "Improved", "No change", or "Worsened". Improved = reduction in WHO FC; No Change = no change in WHO FC; Worsened = increase in WHO FC. The change from baseline in the percentage of participants who improve or show maintenance in WHO FC will be reported.
Change From Baseline in Pulmonary Vascular Resistance (PVR) | Baseline and up to approximately 48 months
  PVR is a hemodynamic variable of pulmonary circulation and is measured by right heart catheterization. The change from baseline in PVR will be reported.
Change From Baseline in Percentage of Participants Who Maintain or Achieve a Low Risk Score Using the Simpliﬁed French Risk Score Calculator | Baseline and up to approximately 48 months
  The simpliﬁed French Risk scoring system is based on the 2015 European Society of Cardiology/European Respiratory Society guidelines for the diagnosis and treatment of pulmonary hypertension (PH). Noninvasive parameters (WHO FC, 6MWD, NT-proBNP levels) will be used to determine the score. 'Low risk' is deﬁned as maintaining or achieving all 3 low-risk criteria: WHO FC I or II, 6MWD >440 meters, and NT-proBNP <300 ng/L. The change from baseline in percentage of participants who maintain or achieve a low risk simpliﬁed French Risk score will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (42):
- United States (14):
  - Pulmonary Associates, PA ( Site 1008), Phoenix, Arizona
  - University of California San Diego Health ( Site 1002), La Jolla, California
  - UCSF Helen Diller Medical Center at Parnassus Heights ( Site 1019), San Francisco, California
  - Jeffrey S. Sager, MD Medical Corporation ( Site 1060), Santa Barbara, California
  - Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center ( Site 1028), Torrance, California
  - University of Colorado Hospital ( Site 1013), Aurora, Colorado
  - Mayo Clinic Jacksonville ( Site 1045), Jacksonville, Florida
  - University of Kansas Medical Center ( Site 1020), Kansas City, Kansas
  - Norton Pulmonary Specialists ( Site 1066), Louisville, Kentucky
  - Tufts Medical Center ( Site 1012), Boston, Massachusetts
  - Weill Cornell Medical Center ( Site 1046), New York, New York
  - The Carl and Edyth Lindner Center for Research and Education at the Christ Hospital ( Site 1001), Cincinnati, Ohio
  - University of Cincinnati Medical Center ( Site 1035), Cincinnati, Ohio
  - Oregon Health & Science University ( Site 1054), Portland, Oregon
- John Hunter Hospital ( Site 1101), New Lambton Heights, New South Wales, Australia
- Vseobecna fakultni nemocnice v Praze ( Site 2201), Prague, Czechia
- Denmark (2):
  - Rigshospitalet ( Site 3802), København Ø, Capital Region
  - Aarhus Universitetshospital, Skejby ( Site 3801), Aarhus, Central Jutland
- France (3):
  - Centre Hospitalier Universitaire de Nice - Hopital Pasteur ( Site 1311), Nice, Alpes-Maritimes
  - CHU Angers ( Site 1313), Angers, Maine-et-Loire
  - Hôpital Louis Pradel ( Site 1317), Lyon, Rhone
- Netherlands (2):
  - Radboud University Nijmegen Medical Centre ( Site 2605), Nijmegen, Gelderland
  - Amsterdam UMC, locatie VUmc ( Site 2601), Amsterdam, North Holland
- Waikato Hospital ( Site 2702), Hamilton, Waikato Region, New Zealand
- South Korea (3):
  - Gachon University Gil Medical Center ( Site 3103), Incheon
  - Severance Hospital, Yonsei University Health System ( Site 3101), Seoul
  - Samsung Medical Center ( Site 3106), Seoul
- Spain (6):
  - Hospital Universitario de Son Espases ( Site 1611), Palma de Mallorca, Balearic Islands
  - Hospital Universitario Marques de Valdecilla ( Site 1601), Santander, Cantabria
  - Hospital Universitario 12 de Octubre ( Site 1603), Madrid, Madrid, Comunidad de
  - Hospital Clinic de Barcelona ( Site 1602), Barcelona
  - Hospital General Universitario Ramon y Cajal ( Site 1609), Madrid
  - HOSPITAL GENERAL UNIVERSITARIO DE TOLEDO ( Site 1607), Toledo
- Sahlgrenska Universitetssjukhuset ( Site 3201), Gothenburg, Västra Götaland County, Sweden
- UniversitätsSpital Zürich ( Site 3301), Zurich, Switzerland
- Taiwan (2):
  - Kaohsiung Veteran General Hospital ( Site 3702), Kaohsiung City
  - National Cheng Kung University Hospital ( Site 3703), Tainan
- United Kingdom (5):
  - Papworth Hospital NHS Foundation Trust ( Site 1208), Cambridge, Cambridgeshire
  - Royal Brompton Hospital ( Site 1206), London, London, City of
  - Hammersmith Hospital ( Site 1203), London, London, City of
  - Freeman Hospital ( Site 1205), Newcastle upon Tyne
  - Royal Hallamshire Hospital ( Site 1207), Sheffield

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- [Result] Preston IR, Badesch D, Ghofrani HA, Gibbs JSR, Gomberg-Maitland M, Hoeper MM, Humbert M, McLaughlin VV, Waxman AB, Manimaran S, Mikhailova E, Reddy M, Lau A, de Oliveira Pena J, Souza R. A long-term follow-up study of sotatercept for treatment of pulmonary arterial hypertension: interim results of SOTERIA. Eur Respir J. 2025 Jul 24;66(1):2401435. doi: 10.1183/13993003.01435-2024. Print 2025 Jul. PMID 39978862
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com